CLINICAL TRIAL: NCT04312230
Title: The Role of Biomarkers in Inherited Cardiac Conditions
Status: Withdrawn | Type: Observational
Why Stopped: Funder has ceased trading and all clinical consultations now held virtually due to COVID
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: ICC-01
Record Dates: First submitted 2019-02-01; First posted 2020-03-18 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Inherited Cardiac Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — As part of this study, all patients due to attend the ICC at USHM will be approached over a 5 year period. The expectation is to recruit 750 patients. Patients will undergo their clinic appointments in the usual manner. As part of the study, a peripheral blood sample of approximately 10mL will be taken to allow measurement of cardiac biomarkers in order to further characterise cardiovascular status and to relate clinical findings to other markers of cardiac disease. Biomarker levels will be related to the presence and severity of cardiovascular disease, at the time of the clinic visit and over subsequent 10 year follow-up, as documented by validated health status questionnaires and information in patients' medical records.
Oversight: Data Monitoring Committee: No

SUMMARY:
Inherited cardiac conditions (ICC) comprise any hereditary condition which may affect cardiac muscle, vasculature, or conductive system. These conditions sometimes present with sudden cardiac death, and may have significant implications for families. Whilst their prevalence may be rare, our understanding of these conditions has increased over the past decade. ICC Clinics aim to improve the diagnosis, treatment and outcomes of these patients.

The NIH has defined a biomarker as "a characteristic that is objectively measured and evaluated as an indicator of normal biological processes, pathogenic processes, or pharmacologic responses to a therapeutic intervention". Biomarkers can indicate disease characteristics, including markers of clinical disease, or indicators of therapeutic response.

This study aims to investigate the utility of biomarkers in a large cohort of patients who are attending the ICC clinic. Biomarkers will be related to the presence and severity of cardiovascular disease and other markers of cardiac disease.

DETAILED DESCRIPTION:
Inherited cardiac conditions (ICC) comprise any hereditary condition which may affect cardiac muscle, vasculature, or conductive system. More than 50 ICCs have been recognised and our diagnostic capabilities ever improve. However, whilst our understanding of ICCs and their molecular basis has increased, management of these conditions remains challenging owing to their heterogeneity, both genetically and clinically. ICC clinics aim to improve and standardise the care of patients with ICCs but improving diagnosis, risk stratification, and management, and by coordinating specialist care provided by other specialities. The UHSM ICC clinic has recently been established, providing tertiary care for patients across a large geographical area. As such, it is well placed is well placed to do this study.

Sudden cardiac death may be the first presentation of ICC, and a new diagnosis has significant implications for families. Risk may be augmented by a multitude of clinical and genetic factors, and there is an increasing need for tools that may be used by clinicians to identify patients at increased risk. Biomarkers are one such tool which may be able to assist in the complex identification of high-risk individuals, to effectively prognosticate and monitor treatment patients with disease.

As part of this study, all patients due to attend the ICC at USHM will be approached over a 5 year period. The expectation is to recruit 750 patients. Patients will undergo their clinic appointments in the usual manner. As part of the study, a peripheral blood sample of approximately 10mL will be taken to allow measurement of cardiac biomarkers in order to further characterise cardiovascular status and to relate clinical findings to other markers of cardiac disease. Biomarker levels will be related to the presence and severity of cardiovascular disease, at the time of the clinic visit and over subsequent 10 year follow-up, as documented by validated health status questionnaires and information in patients' medical records.

This is an observational study of patients referred clinically to the Inherited Cardiac Conditions clinic at the University Hospital of South Manchester.

As part of this study, all patients referred to this clinic will be approached over a 5 year period. The expectation is to recruit 150 patient per year.Patients will attend clinic and other related clinically indicated appointments in the usual manner. As part of the study, a blood sample of approximately 10mL will be taken from the patients arm to allow measurement of cardiac biomarkers in order to further characterise cardiovascular status and to relate these findings to other markers of cardiac disease.

The patient will also be asked to complete a questionnaire about their symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient attending the inherited cardiac conditions clinic

Exclusion Criteria:

* Age < 16 years, Imprisonment Inability to provide informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is an observational study of patients referred clinically to the Inherited Cardiac Conditions clinic at the University Hospital of South Manchester. As part of this study, all patients referred to this clinic will beapproached over a 5 year period. The expectation is to recruit 150 patient per year.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
To establish to role of biomarkers in inherited cardiac conditions | 5 years
  Biomarker profile of patients with cardiomyopathy. Describe the circulating biomarker characteristics of patients with cardiomyopathy, including troponin

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Miller, MBChB PhD, Principal Investigator — Manchester University NHS FT
Locations (1):
- MFT, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT04312230/Prot_SAP_000.pdf